CLINICAL TRIAL: NCT04911335
Title: Sicurezza ed Efficacia di un Prodotto a Base di Propoli (FARINGEL PLUS) Nella Prevenzione e Nel Trattamento Della Mucosite Orale in Pazienti in Cure Palliative: Uno Studio di Fase 2
Brief Title: Propolis-based Product (FARINGEL PLUS) for Oral Mucositis in Palliative Care
Acronym: FARINGEL-CP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Michela Piredda, Associate Professor, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.82
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Oral Mucositis
Keywords: Palliative care; Hospice; Home palliative care; Oral assessment guide
MeSH Terms: conditions — Stomatitis | interventions — faringel; Oral Hygiene

STUDY DESIGN:
Intervention Model Description: Two-step design according to Simon's Optimum approach (1989). Overall sample = 77 evaluable cases (step1_26 cases; step2_51 cases). Parameters: P0 (minimum probability of response): 0.45; P1 (probability of optimal response): 0.60; Alpha: 5%; Power: 80%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phase 2 open intervention (Experimental): All patients assisted by the palliative care center (hospice and home) will receive the oral hygiene protocol and the propolis-based product. The oral hygiene protocol will be applied starting from the day of taking care of the patient in the service and until discharge / death. Administration of the study product will be continued for 2 weeks or stopped sooner if the patient loses the ability to swallow.
  Interventions: Combination Product: Faringel plus and oral hygiene

INTERVENTIONS:
Combination Product: Faringel plus and oral hygiene — The expected frequency of administration of the study product is 2 / day, 10 minutes 'before main meals, for patients without mucositis (grade 1 according to the OAG scale, total score = 8). The frequency of administration will increase to 3 / day for patients with mild or moderate mucositis (grade 2 on the OAG scale, total score 9-18) and up to 4 / day in cases of severe mucositis (grade 3 on the OAG scale, score total 19-24). Each administration will contain 7 ml of oral suspension, to be kept inside the oral cavity for 1-2 minutes and then swallowed slowly.

SUMMARY:
Oral health is crucial for palliative patients' quality of life. The evidence on effective interventions and measures of oral mucositis in palliative care is sparse.

This is a single-center, prospective, uncontrolled open label Phase 2 non-profit study, aimed at evaluating a propolis-based product (FARINGEL PLUS) added to basic oral hygiene safety, acceptability and activity in preventing and treating oral mucositis in patients in palliative care.

A two-step design was adopted according to Simon's Optimum approach, with an overall sample of 77 evaluable cases (step1_26 cases; step2_51 cases).

DETAILED DESCRIPTION:
Palliative Care with has primary objective of the best possible quality of life for patients with advanced illness. Oral health is crucial for quality of life. Oral disorders such as hyposalivation, mucositis, erythema, ulceration and viral and fungal infections, can cause annoying symptoms such as dry mouth, dysphagia, dysgeusia, orofacial pain and speech difficulties, which negatively affect nutrition, verbal communication, social interaction and sleep. An Italian study of advanced cancer patients in palliative care found a prevalence of oral mucositis of 22%, of dysphagia of 15% and of dry mouth of 40%.

Studies on interventions aimed at preventing and treating oral mucositis in palliative care are scarse and no standard oral protocol can be recommended.

Moreover, there are no known scales specifically developed and validated for the evaluation of mucositis and other disorders of the oral cavity in palliative care.

Propolis has historically been used as folk medicine due to multiple biological properties, such as anesthetic, antimicrobial, antifungal, antiviral, and anti-inflammatory for the oral and pharyngeal mucosa. Propolis is effective in reducing the severity of radiation-induced oral mucositis in animals, is associated with a significant reduction in the number and size of oral ulcers in patients diagnosed with recurrent stomatitis and with complete recovery from denture-related stomatitis, and is found safe, acceptable and with promising efficacy in preventing oral mucositis in patients undergoing chemotherapy for breast cancer.

In particular, an oral suspension based on propolis (Faringel) and containing aloe vera gel, calendula, chamomile and sodium alginate, has been found to be well accepted, safe and promising in the prevention of severe oesophagitis from radiotherapy in patients with lung cancer. Hyaluronic acid (Faringel plus) has recently been added to this suspension with a re-epithelizing function on the mucous membranes.

Therefore, we planned this single-center, prospective, uncontrolled open label Phase 2 non-profit study aimed at evaluating whether the addition of a propolis-based product (FARINGEL PLUS) to a basic oral hygiene protocol can be safe, acceptable and active in the protection of the oral cavity in patients in palliative care.

To verify this hypothesis, a two-step design was adopted according to Simon's Optimum design approach. An overall sample of 77 evaluable cases was defined (step1_26 cases; step2_51 cases).

ELIGIBILITY:
Inclusion Criteria:

* Patients cared for by specialized palliative care center in hospice or at home
* Conscious patients able to swallow (score 1-2 at the swallowing item of OAG)
* Patients with a life expectancy of between one week and one month estimated with the RAD (Approximation of Death Recognition) card in use in the palliative care center where the study will be conducted;
* Patients who provide consent to participate in the study and use the data independently, or through their legal representative.

Exclusion Criteria:

* Patients with a life expectancy of less than one week or more than one month estimated with the RAD (Approximation of Death Recognition) card;
* Patients who are unable to swallow (score 3 on the swallowing item on the OAG scale)
* Patients with head / neck cancer or tracheostomy;
* Patients who report allergy to propolis, honey, aloe, chamomile, calendula, stevia (or other components of the product under study) or atopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Severity of oral mucositis | daily up to 15 days
  Reduction of the severity of mucositis by at least one degree, or maintenance of the normal condition, measured by the elements of the OAG scale whose score indicates 3 degrees (from 1 normal condition to 3 severe mucositis). The minimum grade achieved during the patient's stay in the study will be considered.

SECONDARY OUTCOMES:
orpharyngeal pain | daily up to 15 days
  Appearance and severity of oropharyngeal pain assessed with a Numerical Rating Scale (NRS), from 0 to 10 meaning 0 the absence of pain and 10 the worst pain imaginable
esophageal pain | daily up to 15 days
  Appearance and severity of esophageal pain assessed with a Numerical Rating Scale (NRS), from 0 to 10 meaning 0 the absence of pain and 10 the worst pain imaginable
dysgeusia | daily up to 15 days
  Dysgeusia assessed with a Numerical Rating Scale (NRS), from 0 to 10 meaning 0 the absence of symptom and 10 the worst symptom imaginable
ability to swallow, voice condition, feeling of dry mouth | daily up to 15 days
  ability to swallow, voice condition, feeling of dry mouth assessed through the Oral Assessment Guide (OAG - Eilers 1988; D'Angelo et al., 2013) at 3 levels of severity (from 1 normal condition, 2 mild disorders / moderate, 3 severe disorders) and the Tardieu scale, at 4 levels of severity, where 0 is normal and 3 is the maximum degree of alteration).
Oral fungal infections | daily up to 15 days
  Presence and severity of fungal infections measured with CTC-AE (grade 0-5)
Duration of oral disorders | daily up to 15 days
  Duration of oral cavity disorders measured in days and defined from the moment in which a degree different from normality occurs until the first evaluation with return to normality;
Comfort during feeding | daily up to 15 days
  Alteration of comfort during feeding measured daily with a Numerical Rating Scale (NRS), from 0 to 10 (0 complete absence of comfort and 10 maximum comfort)
Meal completion rate | daily up to 15 days
  Food pattern compared to that of the 3 previous days and to the normal situation, measured in number of meals per day and average percentage of completion of individual meals
Patient quality of life | Every 3 days up to 15 days
  Quality of life measured at time 0 and then every 3 days with the European Quality of Life Utility Scale (EQ-5D)
Patient oral-related quality of life | Daily up to 15 days
  Oral-related quality of life measured with the Oral Mucositis Daily Questionnaire (OMDQ)
Adherence to intervention | daily up to 15 days
  Adherence to oral care and to administration of the product under study recorded daily as frequency, type and quantity

CONTACTS AND LOCATIONS:
Overall Officials: Michela Piredda, Dr, Principal Investigator — Campus BioMedico di Roma University
Locations (1):
- Centro di cure palliative Insieme per la cura, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all the IPD that undely a publication, after the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end of the study, and for 3 years after publication of results
Access Criteria: Investigators registered on Clinical.trial.gov who require the data

REFERENCES:
- [Background] Magnani C, Mastroianni C, Giannarelli D, Stefanelli MC, Di Cienzo V, Valerioti T, Casale G. Oral Hygiene Care in Patients With Advanced Disease: An Essential Measure to Improve Oral Cavity Conditions and Symptom Management. Am J Hosp Palliat Care. 2019 Sep;36(9):815-819. doi: 10.1177/1049909119829411. Epub 2019 Feb 12. PMID 30754984
- [Background] Mercadante S, Aielli F, Adile C, Ferrera P, Valle A, Fusco F, Caruselli A, Cartoni C, Massimo P, Masedu F, Valenti M, Porzio G. Prevalence of oral mucositis, dry mouth, and dysphagia in advanced cancer patients. Support Care Cancer. 2015 Nov;23(11):3249-55. doi: 10.1007/s00520-015-2720-y. Epub 2015 Apr 3. PMID 25832897
- [Background] Piredda M, Facchinetti G, Biagioli V, Giannarelli D, Armento G, Tonini G, De Marinis MG. Propolis in the prevention of oral mucositis in breast cancer patients receiving adjuvant chemotherapy: A pilot randomised controlled trial. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12757. Epub 2017 Aug 25. PMID 28840622
- [Derived] Mastroianni C, Marchetti A, Sguanci M, Amato S, Giannarelli D, Casale G, Piredda M, De Marinis MG. Concordance of the World Health Organization, Oral Assessment Guide, and Tardieu Scales for Assessment of Oral Mucositis and Oral Disorders in Palliative Care Patients. J Palliat Med. 2025 Sep;28(9):1239-1245. doi: 10.1089/jpm.2024.0505. Epub 2025 Apr 8. PMID 40197962
- [Derived] Piredda M, Mastroianni C, Marchetti A, Sguanci M, Farinella R, Natale M, Giannarelli D, Monaco E, Martinato M, Armento G, Casale G, De Marinis MG. A Propolis-Based Protocol for Oral Health in Palliative Care: Results from a Phase II Trial. J Palliat Med. 2025 Feb;28(2):243-250. doi: 10.1089/jpm.2024.0290. Epub 2024 Dec 23. PMID 39711194